CLINICAL TRIAL: NCT04010539
Title: A Phase III, Randomized, Multicenter, Open-Label Study in Adolescent and Adult Participants Comparing the Efficacy and Safety of Gepotidacin to Ceftriaxone Plus Azithromycin in the Treatment of Uncomplicated Urogenital Gonorrhea Caused by Neisseria Gonorrhoeae
Brief Title: A Study Evaluating Efficacy and Safety of Gepotidacin Compared With Ceftriaxone Plus Azithromycin in the Treatment of Uncomplicated Urogenital Gonorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116577; 2018-001780-23 (EudraCT Number)
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-04

CONDITIONS: Gonorrhea
Keywords: Urogenital Gonorrhea; Gepotidacin; Neisseria gonorrhoeae; Efficacy; Phase 3
MeSH Terms: conditions — Gonorrhea | interventions — gepotidacin; Ceftriaxone; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving Gepotidacin (Experimental): Participants will receive Gepotidacin orally at the study site during the Baseline (Day 1) visit followed by self-administration of a second oral dose as an outpatient 10 to 12 hours after the first dose.
  Interventions: Drug: Gepotidacin
- Participants receiving Ceftriaxone plus Azithromycin (Active Comparator): Participants will receive a single IM dose of Ceftriaxone plus a single oral dose of Azithromycin at the study site during the Baseline (Day 1) visit.
  Interventions: Drug: Ceftriaxone; Drug: Azithromycin

INTERVENTIONS:
Drug: Gepotidacin — Gepotidacin will be administered as 3000 milligram (mg) oral dose (4 X 750 mg tablets) at the study site followed by 3000 mg oral dose (4 X 750 mg tablets) as an outpatient. Each dose should be taken after food consumption and with water.
  Arms: Participants receiving Gepotidacin
Drug: Ceftriaxone — Ceftriaxone is available as sterile powder for reconstitution. It will be administered as one 500-mg IM dose at the study site.
  Arms: Participants receiving Ceftriaxone plus Azithromycin
Drug: Azithromycin — Azithromycin will be administered as 1000 mg oral dose (2 X 500 mg tablets) at the study site. Dose should be taken after food consumption and with water.
  Arms: Participants receiving Ceftriaxone plus Azithromycin

SUMMARY:
This is a phase III, randomized, multicenter, open-label study which will be performed to evaluate efficacy and safety of oral Gepotidacin compared to intramuscular (IM) ceftriaxone plus oral azithromycin for the treatment of uncomplicated urogenital infection caused by Neisseria gonorrhoeae (N. gonorrhoeae) in adolescent and adult participants. In this study, participants will be randomly assigned to receive either oral gepotidacin or IM ceftriaxone plus oral azithromycin.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be >=12 years of age at the time of signing the informed consent.
* Participants having body weight of >45 kilogram (kg).
* Participants having clinical suspicion of a urogenital gonococcal infection with or without pharyngeal and/or rectal gonococcal infection and have one of the following: male participants with purulent yellow, green, or white urethral discharge or female participants with abnormal cervical or vaginal mucopurulent discharge upon physical examination; or a prior positive culture for N. gonorrhoeae from up to 5 days before screening (as long as the participant has not received any treatment for this infection); or a Gram or equivalent stain (urogenital specimens only) positive or presumptive for Gram-negative intracellular diplococci from up to 5 days before screening (as long as the participant has not received any treatment for this infection); or a prior positive nucleic acid amplification test assay for N. gonorrhoeae from up to 7 days before screening (as long as the participant has not received any treatment for this infection).
* Participants who are willing to avoid anal, oral, and vaginal sexual intercourse or use condoms for all forms of intercourse from the Baseline Visit through the TOC Visit.
* Male or female participants having his or her original urogenital anatomy at birth.
* Male participant must agree to use contraception (male condoms) during intercourse from the Baseline Visit through completion of the TOC Visit.
* Female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies: Not a woman of childbearing potential (WOCBP) or WOCBP who agrees to follow the contraceptive guidance (male partners of WOCBP must use a male condom during intercourse) from the Baseline Visit through completion of the TOC Visit.
* Participants who are capable of giving signed informed consent or assent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) or assent form and in study protocol.

Exclusion Criteria:

* Male participants with a current diagnosis of epididymitis and/or orchitis at the time of the Baseline Visit.
* Participant who is suspected or confirmed to have a Chlamydia trachomatis infection and per the investigator's judgement standard-of-care treatment for this infection cannot be safely postponed until the TOC Visit.
* Participant has a body mass index >=40 kilogram per square meter (kg/m^2) or has a body mass index >=35.0 kg/m^2 and is experiencing obesity-related health conditions such as high blood pressure or diabetes.
* Participant has a history of sensitivity to the study treatments, or components thereof, or a history of a drug (including erythromycin and any macrolide or ketolide drug) or other allergy that, in the opinion of the investigator or medical monitor, contraindicates his or her participation.
* Participant is immunocompromised or has altered immune defenses that may predispose the participant to a higher risk of treatment failure and/or complications.
* Participants with a known cluster of differentiation 4 (CD4) count of <200 cells per cubic millimeter (cells/mm^3).
* Participant has any of the following: poorly controlled asthma or chronic obstructive pulmonary disease, acute severe pain, uncontrolled with conventional medical management, active peptic ulcer disease, Parkinson disease, Myasthenia gravis, a history of seizure disorder requiring medications for control or participant has any surgical or medical condition that may interfere with drug absorption, distribution, metabolism, or excretion of the study treatment.
* Participant has known anuria, oliguria, or severe impairment of renal function (creatinine clearance <30 milliliter per minute [mL/min] or clinically significant elevated serum creatinine as determined by the investigator).
* Participant in the judgment of the investigator, would not be able or willing to comply with the protocol or complete study follow-up.
* Participant has a serious underlying disease that could be imminently life threatening, or the participant is unlikely to survive for the duration of the study period.
* Participant has congenital long QT syndrome or known prolongation of corrected QT interval (QTc).
* Participant has uncompensated heart failure.
* Participant has severe left ventricular hypertrophy.
* Participant has a family history of QT prolongation or sudden death.
* Participant has a recent history of vasovagal syncope or episodes of symptomatic bradycardia or bradyarrhythmia within the last 12 months.
* The participant is taking QT-prolonging drugs or drugs known to increase the risk of torsades de pointes (TdP) per the www.crediblemeds.org "Known Risk of TdP" category at the time of his or her Baseline Visit, which cannot be safely discontinued from the Baseline Visit to the TOC Visit; or the participant is taking a strong cytochrome P450 enzyme 3A4 (CYP3A4) inhibitor or a strong P-glycoprotein (P-gp) inhibitor.
* For any participant >=12 to <18 years, the participant has an abnormal electrocardiogram (ECG) reading.
* The participant has a QTc >450 millisecond (msec) or a QTc >480 msec for participants with bundle-branch block.
* Participant has a documented or recent history of uncorrected hypokalemia within the past 3 months.
* Participant has a known history of cholestatic jaundice or hepatic dysfunction associated with prior use of azithromycin.
* Participant has a known alanine aminotransferase (ALT) value >2 times upper limit of normal (ULN).
* Participant has a known bilirubin value >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Participant has a current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), including symptomatic viral hepatitis or moderate-to-severe liver insufficiency (Child Pugh class B or C).
* Participant has been previously randomized in this study or has previously been treated with Gepotidacin.
* Participant has participated in a clinical trial and has received an investigational product within 30 days or 5 half-lives, whichever is longer.
* Participant has any of the following gonococcal infections that require a different dose or duration of treatment: suspected or confirmed pelvic inflammatory disease; or suspected or confirmed gonococcal arthritis; or suspected or confirmed gonococcal conjunctivitis; or suspected or confirmed gonococcal endocarditis; or other evidence of disseminated gonococcal infection.
* Participant has received any antibacterial therapy for the treatment of a gonococcal infection within 14 days before the Baseline Visit.
* Participant has received any systemic, topical, or intravaginal antibiotics or any systemic antifungals within 7 days before the Baseline Visit.
* Participant must not use St John's wort or ergot derivatives from within 14 days before the Baseline Visit through the TOC Visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (38):
- United States (13):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
- Australia (5):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Darlinghurst, Sydney, New South Wales
  - GSK Investigational Site, Southport, Queensland
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Prahran, Victoria
- Germany (6):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, München
- Mexico (2):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville
- United Kingdom (8):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Brighton
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Reading
  - GSK Investigational Site, St Helens

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

REFERENCES:
- [Derived] Ross JDC, Wilson J, Workowski KA, Taylor SN, Lewis DA, Gatsi S, Flight W, Scangarella-Oman NE, Jakielaszek C, Lythgoe D, Powell M, Janmohamed S, Absalon J, Perry C. Oral gepotidacin for the treatment of uncomplicated urogenital gonorrhoea (EAGLE-1): a phase 3 randomised, open-label, non-inferiority, multicentre study. Lancet. 2025 May 3;405(10489):1608-1620. doi: 10.1016/S0140-6736(25)00628-2. Epub 2025 Apr 14. PMID 40245902
- [Derived] Perry CR, Scangarella-Oman NE, Millns H, Flight W, Gatsi S, Jakielaszek C, Janmohamed S, Lewis DA. Efficacy and Safety of Gepotidacin as Treatment of Uncomplicated Urogenital Gonorrhea (EAGLE-1): Design of a Randomized, Comparator-Controlled, Phase 3 Study. Infect Dis Ther. 2023 Sep;12(9):2307-2320. doi: 10.1007/s40121-023-00862-6. Epub 2023 Sep 26. PMID 37751016
- [Derived] Fishman C, Caverly Rae JM, Posobiec LM, Laffan SB, Lerman SA, Pearson N, Janmohamed S, Dumont E, Nunn-Floyd D, Stanislaus DJ. Novel Bacterial Topoisomerase Inhibitor Gepotidacin Demonstrates Absence of Fluoroquinolone-Like Arthropathy in Juvenile Rats. Antimicrob Agents Chemother. 2022 Nov 15;66(11):e0048322. doi: 10.1128/aac.00483-22. Epub 2022 Oct 18. PMID 36255258

RESULTS

PARTICIPANT FLOW:
Groups:
- Gepotidacin: Participants with uncomplicated urogenital gonorrhea (GC) were randomized to receive first dose of 3000 milligram (mg) (4*750 mg, tablets) gepotidacin orally on Day 1. Participants self-administered second dose of 3000 mg (4*750 mg, tablets) gepotidacin orally 10-12 hours after first dose. All doses were to be administered after food consumption and with water.
- Ceftriaxone Plus Azithromycin: Participants with uncomplicated urogenital gonorrhea (GC) were randomized to receive single dose of 500 mg Ceftriaxone as intramuscular sterile powder reconstituted with appropriate diluent plus single oral dose of 1 gram (g) Azithromycin (2*500 mg, tablets) on Day 1. Azithromycin was to be administered after food consumption and with water.
Period: Overall Study
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Started (Intent-to-Treat (ITT) Population: All participants randomly assigned to study treatment.) | 314 | 314
Safety Population (All participants who received at least 1 dose of study treatment.) | 309 | 313
Microbiological ITT (Micro-ITT) Population (All participants randomly assigned to study treatment who received at least 1 dose of study treatment and have confirmed NG isolated that is ceftriaxone-susceptible (based on Clinical & Laboratory Standards Institute (CLSI) breakpoints) from baseline culture of their urogenital specimen.) | 202 | 204
Micro-ITT Rectal Population (All participants who met the definition of the Micro-ITT Population and have confirmed NG isolated that is ceftriaxone-susceptible (based on CLSI breakpoints) from baseline culture of their rectal specimen.) | 26 | 15
Micro-ITT Pharyngeal Population (All participants who met the definition of the Micro-ITT Population and have confirmed NG isolated that is ceftriaxone-susceptible (based on CLSI breakpoints) from baseline culture of their pharyngeal specimen.) | 18 | 17
Completed | 294 | 295
Not Completed | 20 | 19
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Lost to Follow-up | 10 | 14
Not completed — Adverse Event | 3 | 0
Not completed — Participant Did Not Receive IP | 0 | 1
Not completed — Protocol Deviation | 0 | 1
Not completed — Randomized in Error/ Mistake | 2 | 0
Not completed — Eligibility Criteria Unable to Evaluate | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin | Total
Number analyzed (Participants) | 314 | 314 | 628
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.9 (10.42) | 33.7 (10.70) | 33.8 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 279 | 280 | 559
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 10 | 19
  Asian | 12 | 17 | 29
  Native Hawaiian or Other Pacific Islander | 7 | 2 | 9
  Black or African American | 49 | 39 | 88
  White | 231 | 241 | 472
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Culture-Confirmed Bacterial Eradication of Neisseria Gonorrhoeae (NG) From the Urogenital Site at the Test-Of-Cure (TOC) Visit (Day 4 to 8)
Description: Urogenital specimens were obtained for bacteriological culture at the Baseline (Day 1) and TOC (Day 4 to 8) visits and were compared to determine microbiological outcome. Microbiological success was defined as culture-confirmed elimination of baseline pathogen (NG) from a bacteriology sample taken at the TOC visit without the participant receiving other systemic antimicrobials before this visit. Microbiological failure was categorized as "Bacterial Persistence (BP)" and "Unable to Determine (UTD)" outcomes. Bacterial persistence was defined as culture-confirmed persistence of baseline NG pathogen from a bacteriology sample taken at the TOC visit without the participant receiving other systemic antimicrobials before this visit. UTD was defined as inability to determine the TOC NG pathogen outcome (e.g., no bacteriological sample taken for culture, sample lost, visit did not occur etc.) or the participant received other systemic antimicrobials before the TOC visit.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Microbiological intent-to-treat (Micro-ITT) population included all participants randomly assigned to study treatment who received at least 1 dose of study treatment and have confirmed NG isolated that is ceftriaxone-susceptible (based on CLSI breakpoints) from baseline culture of their urogenital specimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 202 | 204
Participants
  Microbiological success | 187 | 186
  Microbiological failure, BP | 0 | 0
  Microbiological failure, UTD | 15 | 18
Statistical Analysis 1: Comparison: Gepotidacin vs Ceftriaxone Plus Azithromycin; Test type: Non-Inferiority — The difference in microbiological success rates between treatment groups (Gepotidacin - Ceftriaxone plus azithromycin) was calculated using the Miettinen-Nurminen Summary Score Method adjusted for sex and sexual orientation combination. Non-inferiority was declared if the lower limit of the 2-sided 95% confidence interval for the difference was above -10.0%; Adjusted Difference in Percent = -0.1, 95% CI 2-sided [-5.6 to 5.5]
Statistical Analysis 2: Comparison: Gepotidacin vs Ceftriaxone Plus Azithromycin; Test type: Superiority — The difference in microbiological success rates between treatment groups (Gepotidacin - Ceftriaxone plus azithromycin) was calculated using the Miettinen-Nurminen Summary Score Method adjusted for sex and sexual orientation combination. Superiority was declared if the lower limit of the 2-sided 95% confidence interval for the difference was above 0.0%; p = 0.5072, 1-sided p-value for Test of Superiority; Adjusted Difference in Percent = -0.1, 95% CI 2-sided [-5.6 to 5.5]

2. Secondary Outcome: Number of Participants With Culture-Confirmed Bacterial Eradication of NG From the Rectal Site at the TOC Visit
Description: Rectal specimens were obtained for bacteriological culture at the Baseline (Day 1) and TOC (Day 4 to 8) visits and were compared to determine microbiological outcome. Microbiological success was defined as culture-confirmed elimination of baseline pathogen (NG) from a bacteriology sample taken at the TOC visit without the participant receiving other systemic antimicrobials before this visit. Microbiological failure was categorized as "Bacterial Persistence (BP)" and "Unable to Determine (UTD)" outcomes. Bacterial persistence was defined as culture-confirmed persistence of baseline NG pathogen from a bacteriology sample taken at the TOC visit without the participant receiving other systemic antimicrobials before this visit. UTD was defined as inability to determine the TOC NG pathogen outcome (e.g., no bacteriological sample taken for culture, sample lost, visit did not occur etc.) or the participant received other systemic antimicrobials before the TOC visit.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Micro-ITT Rectal population included all participants who met the definition of the Micro-ITT Population and have confirmed NG isolated that is ceftriaxone susceptible from baseline culture of their rectal specimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 26 | 15
Participants
  Microbiological success | 26 | 12
  Microbiological failure, BP | 0 | 0
  Microbiological failure, UTD | 0 | 3

3. Secondary Outcome: Number of Participants With Culture-Confirmed Bacterial Eradication of NG From the Pharyngeal Site at the TOC Visit
Description: Pharyngeal specimens were obtained for bacteriological culture at the Baseline (Day 1) and TOC (Day 4 to 8) visits and were compared to determine microbiological outcome. Microbiological success was defined as culture-confirmed elimination of baseline pathogen (NG) from a bacteriology sample taken at the TOC visit without the participant receiving other systemic antimicrobials before this visit. Microbiological failure was categorized as "Bacterial Persistence (BP)" and "Unable to Determine (UTD)" outcomes. Bacterial persistence was defined as culture-confirmed persistence of baseline NG pathogen from a bacteriology sample taken at the TOC visit without the participant receiving other systemic antimicrobials before this visit. UTD was defined as inability to determine the TOC NG pathogen outcome (e.g., no bacteriological sample taken for culture, sample lost, visit did not occur etc.) or the participant received other systemic antimicrobials before the TOC visit.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Micro-ITT Pharyngeal population included all participants who met the definition of the Micro-ITT Population and have confirmed NG isolated that is ceftriaxone susceptible from baseline culture of their pharyngeal specimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 18 | 17
Participants
  Microbiological success | 14 | 16
  Microbiological failure, BP | 2 | 0
  Microbiological failure, UTD | 2 | 1

4. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs) and Any Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A TEAE is an event that emerges during treatment having been absent pretreatment or worsens relative to the pretreatment state. An SAE is defined as any untoward medical occurrence that, at any dose, results in death; was life threatening; required hospitalization or prolongation of existing hospitalization; resulted in disability/incapacity; was a congenital anomaly/birth defect.
Time Frame: Up to 21 days
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 309 | 313
Participants
  Any TEAEs | 230 | 104
  Any SAEs | 1 | 0

5. Secondary Outcome: Change From Baseline (CFB) in Hematology Parameters: Basophils, Eosinophil, Leukocytes, Neutrophils, Platelets, Lymphocytes, Monocytes, Neutrophils and Nucleated Erythrocytes
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters: basophils, eosinophil, leukocytes, neutrophils, platelets, lymphocytes, monocytes, neutrophils and nucleated erythrocytes. Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9 cells/L)
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 284 | 293
Giga cells per liter (10^9 cells/L)
  Basophils, Baseline (Day 1) | 0.044 (0.0196) | 0.045 (0.0222)
  Basophils, CFB to TOC: number analyzed (Participants) | 256 | 268
  Basophils, CFB to TOC | 0.001 (0.0167) | 0.000 (0.0152)
  Eosinophils, Baseline (Day 1) | 0.154 (0.2117) | 0.160 (0.1384)
  Eosinophils, CFB to TOC: number analyzed (Participants) | 256 | 268
  Eosinophils, CFB to TOC | 0.009 (0.1289) | 0.018 (0.0827)
  Leukocytes, Baseline (Day 1) | 7.143 (2.2808) | 7.507 (2.2045)
  Leukocytes, CFB to TOC: number analyzed (Participants) | 256 | 268
  Leukocytes, CFB to TOC | -0.811 (1.8536) | -1.267 (1.9362)
  Neutrophils, Baseline (Day 1) | 4.443 (1.9621) | 4.774 (1.9355)
  Neutrophils, CFB to TOC: number analyzed (Participants) | 256 | 268
  Neutrophils, CFB to TOC | -1.062 (1.7309) | -1.473 (1.8860)
  Platelets, Baseline (Day 1): number analyzed (Participants) | 284 | 290
  Platelets, Baseline (Day 1) | 260.3 (61.79) | 268.4 (69.26)
  Platelets, CFB to TOC: number analyzed (Participants) | 256 | 264
  Platelets, CFB to TOC | 10.2 (32.14) | 9.7 (34.94)
  Lymphocytes, Baseline (Day 1) | 1.934 (0.5941) | 1.948 (0.6321)
  Lymphocytes, CFB to TOC: number analyzed (Participants) | 256 | 268
  Lymphocytes, CFB to TOC | 0.277 (0.5205) | 0.245 (0.5511)
  Monocytes, Baseline (Day 1) | 0.559 (0.2209) | 0.572 (0.1877)
  Monocytes, CFB to TOC: number analyzed (Participants) | 256 | 268
  Monocytes, CFB to TOC | -0.034 (0.1917) | -0.053 (0.1782)
  Nucleated Erythrocytes, Baseline (Day 1): number analyzed (Participants) | 284 | 292
  Nucleated Erythrocytes, Baseline (Day 1) | 0.002 (0.0047) | 0.001 (0.0038)
  Nucleated Erythrocytes, CFB to TOC: number analyzed (Participants) | 256 | 267
  Nucleated Erythrocytes, CFB to TOC | 0.000 (0.0070) | 0.001 (0.0059)

6. Secondary Outcome: Change From Baseline in Hematology Parameters: Mean Corpuscular Hemoglobin Concentration (MCHC) and Hemoglobin (Hb)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters: mean corpuscular hemoglobin concentration and hemoglobin. Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 284 | 293
Grams per liter (g/L)
  MCHC, Baseline (Day 1) | 318.5 (16.27) | 318.8 (16.12)
  MCHC, CFB to TOC: number analyzed (Participants) | 256 | 268
  MCHC, CFB to TOC | 2.4 (10.67) | 0.3 (11.27)
  Hb, Baseline (Day 1) | 149.1 (12.83) | 149.2 (12.58)
  Hb, CFB to TOC: number analyzed (Participants) | 256 | 268
  Hb, CFB to TOC | 0.00 (6.70) | 0.6 (6.92)

7. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter: hematocrit. Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 284 | 293
Percentage
  Baseline (Day 1) | 0.4691 (0.04205) | 0.4687 (0.04104)
  CFB to TOC: number analyzed (Participants) | 256 | 268
  CFB to TOC | -0.0038 (0.02526) | 0.0012 (0.02666)

8. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter: red blood cell (RBC) count. Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter (10^12 cells/L)
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 284 | 293
Trillion cells per liter (10^12 cells/L)
  Baseline (Day 1) | 4.911 (0.4722) | 4.926 (0.4601)
  CFB to TOC: number analyzed (Participants) | 256 | 268
  CFB to TOC | 0.003 (0.2261) | 0.019 (0.2332)

9. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter: mean corpuscular hemoglobin (MCH). Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Picograms (pg)
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 284 | 293
Picograms (pg)
  Baseline (Day 1) | 30.46 (1.978) | 30.38 (1.987)
  CFB to TOC: number analyzed (Participants) | 256 | 268
  CFB to TOC | -0.03 (0.451) | 0.00 (0.594)

10. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Volume (MCV)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter: mean corpuscular volume (MCV). Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters (fL)
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 284 | 293
Femtoliters (fL)
  Baseline (Day 1) | 95.79 (6.266) | 95.43 (6.760)
  CFB to TOC: number analyzed (Participants) | 256 | 268
  CFB to TOC | -0.85 (3.104) | -0.12 (3.084)

11. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Urea Nitrogen (UN), Glucose, Calcium, Chloride, Sodium, Magnesium and Potassium
Description: Blood samples were collected for the assessment of change from baseline in clinincal chemistry parameters: urea nitrogen (UN), glucose, calcium, chloride, sodium, magnesium and potassium. Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 304 | 306
Millimoles per liter (mmol/L)
  UN, Baseline (Day 1): number analyzed (Participants) | 303 | 305
  UN, Baseline (Day 1) | 4.793 (1.4293) | 4.800 (1.4669)
  UN, CFB to TOC: number analyzed (Participants) | 285 | 282
  UN, CFB to TOC | 0.190 (1.1640) | 0.282 (1.1920)
  Glucose, Baseline: number analyzed (Participants) | 298 | 302
  Glucose, Baseline | 5.049 (1.0557) | 5.090 (1.1183)
  Glucose, CFB to TOC: number analyzed (Participants) | 279 | 278
  Glucose, CFB to TOC | 0.227 (0.9425) | 0.064 (0.9684)
  Calcium, Baseline (Day 1): number analyzed (Participants) | 303 | 305
  Calcium, Baseline (Day 1) | 2.387 (0.0986) | 2.387 (0.0954)
  Calcium, CFB to TOC: number analyzed (Participants) | 285 | 282
  Calcium, CFB to TOC | -0.009 (0.0852) | -0.015 (0.0871)
  Chloride, Baseline (Day 1): number analyzed (Participants) | 303 | 305
  Chloride, Baseline (Day 1) | 101.7 (2.26) | 101.7 (2.30)
  Chloride, CFB to TOC: number analyzed (Participants) | 285 | 282
  Chloride, CFB to TOC | 0.7 (2.57) | 0.5 (2.40)
  Sodium, Baseline (Day 1) | 139.6 (2.11) | 139.6 (2.02)
  Sodium, CFB to TOC: number analyzed (Participants) | 286 | 283
  Sodium, CFB to TOC | 0.2 (2.19) | 0.1 (2.44)
  Magnesium, Baseline (Day 1): number analyzed (Participants) | 303 | 305
  Magnesium, Baseline (Day 1) | 0.854 (0.0612) | 0.855 (0.0637)
  Magnesium, CFB to TOC: number analyzed (Participants) | 285 | 282
  Magnesium, CFB to TOC | -0.003 (0.0604) | -0.004 (0.0584)
  Potassium, Baseline (Day 1): number analyzed (Participants) | 300 | 303
  Potassium, Baseline (Day 1) | 4.29 (0.323) | 4.30 (0.332)
  Potassium, CFB to TOC: number analyzed (Participants) | 281 | 278
  Potassium, CFB to TOC | -0.04 (0.336) | -0.03 (0.345)

12. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples were collected for the assessment of change from baseline in clinical chemistry parameters: bilirubin, direct bilirubin and creatinine levels. Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 303 | 305
Micromoles per liter (umol/L)
  Bilirubin, Baseline (Day 1): number analyzed (Participants) | 301 | 304
  Bilirubin, Baseline (Day 1) | 8.54 (5.861) | 7.71 (4.806)
  Bilirubin, CFB to TOC: number analyzed (Participants) | 282 | 280
  Bilirubin, CFB to TOC | -0.05 (5.025) | -0.14 (3.914)
  Direct Bilirubin, Baseline (Day 1): number analyzed (Participants) | 301 | 304
  Direct Bilirubin, Baseline (Day 1) | 3.83 (1.248) | 3.76 (1.210)
  Direct Bilirubin, CFB to TOC: number analyzed (Participants) | 282 | 280
  Direct Bilirubin, CFB to TOC | -0.02 (0.897) | 0.01 (0.876)
  Creatinine, Baseline (Day 1) | 75.9 (34.12) | 75.0 (20.63)
  Creatinine, CFB to TOC: number analyzed (Participants) | 285 | 282
  Creatinine, CFB to TOC | -0.2 (34.08) | 2.6 (9.52)

13. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Albumin and Protein
Description: Blood samples were collected for the assessment of change from baseline in clinical chemistry parameters: albumin and protein. Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 305 | 306
Grams per liter (g/L)
  Albumin, Baseline (Day 1) | 46.9 (3.12) | 46.8 (3.19)
  Albumin, CFB to TOC: number analyzed (Participants) | 287 | 283
  Albumin, CFB to TOC | -0.3 (2.35) | -0.3 (2.67)
  Protein, Baseline (Day 1): number analyzed (Participants) | 301 | 304
  Protein, Baseline (Day 1) | 73.1 (4.80) | 73.3 (4.85)
  Protein, CFB to TOC: number analyzed (Participants) | 282 | 280
  Protein, CFB to TOC | -0.5 (3.86) | -0.5 (4.02)

14. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Alkaline Phosphatase (ALP)
Description: Blood samples were collected for the assessment of change from baseline in clinincal chemistry parameters: aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP). Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter (IU/L)
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 303 | 305
International units per Liter (IU/L)
  AST, Baseline (Day 1): number analyzed (Participants) | 301 | 304
  AST, Baseline (Day 1) | 24.4 (15.30) | 24.2 (16.29)
  AST, CFB to TOC: number analyzed (Participants) | 280 | 280
  AST, CFB to TOC | 2.8 (19.51) | 0.9 (13.25)
  ALT, Baseline (Day 1): number analyzed (Participants) | 301 | 304
  ALT, Baseline (Day 1) | 23.7 (18.78) | 23.7 (14.35)
  ALT, CFB to TOC: number analyzed (Participants) | 281 | 280
  ALT, CFB to TOC | 1.4 (12.59) | 1.1 (7.64)
  ALP, Baseline (Day 1) | 76.0 (20.86) | 77.1 (26.53)
  ALP, CFB to TOC: number analyzed (Participants) | 285 | 282
  ALP, CFB to TOC | -0.4 (7.73) | -1.5 (7.80)

15. Secondary Outcome: Number of Participants With Urinalysis Dipstick Results
Description: Urine samples were collected for urinalysis: Glucose, Protein, Occult Blood and Ketones. The dipstick test gives results in a semi-quantitative manner, and results can be read as Negative, Small, Moderate, Large, Positive, 5 milligram per deciliter (mg/dL), 20 mg/dL, 30 mg/dL 50 mg/dL, 100 mg/dL, 150 mg/dL and >=500 mg/dL indicating concentrations in the urine sample. In the row title (Glucose, Baseline, Negative), Glucose indicates parameter, Baseline is the visit and Negative indicates the concentration in the urine sample. Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 299 | 307
Participants
  Glucose, Baseline (Day 1), Negative | 296 | 305
  Glucose, Baseline (Day 1), 150 mg/dL | 0 | 0
  Glucose, Baseline (Day 1), >=500 mg/dL | 3 | 2
  Glucose, TOC, Negative: number analyzed (Participants) | 287 | 285
  Glucose, TOC, Negative | 284 | 283
  Glucose, TOC, 150 mg/dL: number analyzed (Participants) | 287 | 285
  Glucose, TOC, 150 mg/dL | 1 | 1
  Glucose, TOC, >=500 mg/dL: number analyzed (Participants) | 287 | 285
  Glucose, TOC, >=500 mg/dL | 2 | 1
  Ketones, Baseline (Day 1), Negative | 288 | 300
  Ketones, Baseline (Day 1), 5 mg/dL | 10 | 7
  Ketones, Baseline (Day 1), 20 mg/dL | 1 | 0
  Ketones, TOC, Negative: number analyzed (Participants) | 287 | 285
  Ketones, TOC, Negative | 279 | 279
  Ketones, TOC, 5 mg/dL: number analyzed (Participants) | 287 | 285
  Ketones, TOC, 5 mg/dL | 7 | 6
  Ketones, TOC, 20 mg/dL: number analyzed (Participants) | 287 | 285
  Ketones, TOC, 20 mg/dL | 1 | 0
  Occult Blood, Baseline (Day 1), Negative | 202 | 192
  Occult Blood, Baseline (Day 1), Small | 77 | 91
  Occult Blood, Baseline (Day 1), Moderate | 18 | 19
  Occult Blood, Baseline (Day 1), Large | 2 | 5
  Occult Blood, TOC, Negative: number analyzed (Participants) | 287 | 285
  Occult Blood, TOC, Negative | 251 | 252
  Occult Blood, TOC, Small: number analyzed (Participants) | 287 | 285
  Occult Blood, TOC, Small | 30 | 24
  Occult Blood, TOC, Moderate: number analyzed (Participants) | 287 | 285
  Occult Blood, TOC, Moderate | 3 | 6
  Occult Blood, TOC, Large: number analyzed (Participants) | 287 | 285
  Occult Blood, TOC, Large | 3 | 3
  Protein, Baseline (Day 1), Negative | 212 | 210
  Protein, Baseline (Day 1), 30 mg/dL | 79 | 83
  Protein, Baseline (Day 1), 100 mg/dL | 8 | 13
  Protein, Baseline (Day 1), >=500 mg/dL | 0 | 1
  Protein, TOC, Negative: number analyzed (Participants) | 287 | 285
  Protein, TOC, Negative | 239 | 244
  Protein, TOC, 30 mg/dL: number analyzed (Participants) | 287 | 285
  Protein, TOC, 30 mg/dL | 46 | 37
  Protein, TOC, 100 mg/dL: number analyzed (Participants) | 287 | 285
  Protein, TOC, 100 mg/dL | 2 | 4
  Protein, TOC, >=500 mg/dL: number analyzed (Participants) | 287 | 285
  Protein, TOC, >=500 mg/dL | 0 | 0

16. Secondary Outcome: Absolute Values in Specific Gravity of Urine
Description: Urine samples were collected from participants to assess urine specific gravity. Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 299 | 307
Ratio
  Baseline (Day 1) | 1.0211 (0.00750) | 1.0207 (0.00747)
  TOC: number analyzed (Participants) | 287 | 284
  TOC | 1.0211 (0.00720) | 1.0216 (0.00748)

17. Secondary Outcome: Absolute Values in Potential of Hydrogen (pH) of Urine
Description: Urine samples were collected from participants to assess urine pH. Baseline (Day 1) was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 299 | 307
pH
  Baseline (Day 1) | 5.6 (0.69) | 5.6 (0.70)
  TOC: number analyzed (Participants) | 287 | 285
  TOC | 5.5 (0.64) | 5.4 (0.62)

18. Secondary Outcome: Change From Baseline in Vital Signs: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in a semi-supine position after 5 minutes rest. Baseline (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 307 | 313
Millimeters of mercury (mmHg)
  SBP, Baseline (Day 1) | 123.9 (13.69) | 125.1 (14.41)
  SBP, CFB to TOC: number analyzed (Participants) | 289 | 292
  SBP, CFB to TOC | -0.4 (12.61) | -0.5 (12.86)
  DBP, Baseline (Day 1) | 76.7 (10.77) | 77.2 (10.50)
  DBP, CFB to TOC: number analyzed (Participants) | 289 | 292
  DBP, CFB to TOC | 0.1 (9.10) | -0.9 (9.54)

19. Secondary Outcome: Change From Baseline in Vital Sign: Pulse Rate
Description: Pulse rate was measured in a semi-supine position after 5 minutes rest. Baseline (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 308 | 313
Beats per minute
  Baseline (Day 1) | 73.0 (12.24) | 72.8 (12.20)
  CFB to TOC: number analyzed (Participants) | 290 | 292
  CFB to TOC | 2.2 (12.44) | 2.4 (12.33)

20. Secondary Outcome: Change From Baseline in Vital Sign: Temperature
Description: Temperature was measured after 5 minutes rest. Baseline (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and TOC visit (Day 4 to 8)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Celsius (C)
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
Number analyzed (Participants) | 306 | 313
Celsius (C)
  Baseline (Day 1) | 36.45 (0.395) | 36.44 (0.457)
  CFB to TOC: number analyzed (Participants) | 289 | 292
  CFB to TOC | -0.03 (0.381) | -0.06 (0.485)

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected from Day 1 through the final follow-up visit (up to 21Days).
Description: Safety population included all participants who received at least 1 dose of study treatment.
Arm/Group | Gepotidacin | Ceftriaxone Plus Azithromycin
All-Cause Mortality (participants affected / at risk) | 0/309 | 0/313
Serious Adverse Events (participants affected / at risk) | 1/309 | 0/313
Other Adverse Events (participants affected / at risk) | 230/309 | 81/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gepotidacin (N=309) | Ceftriaxone Plus Azithromycin (N=313)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gepotidacin (N=309) | Ceftriaxone Plus Azithromycin (N=313)
Diarrhoea (Gastrointestinal disorders) | 151 (167) | 30 (30)
Nausea (Gastrointestinal disorders) | 73 (80) | 9 (9)
Vomiting (Gastrointestinal disorders) | 20 (21) | 2 (2)
Flatulence (Gastrointestinal disorders) | 20 (20) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 16 (17) | 3 (4)
Faeces soft (Gastrointestinal disorders) | 16 (16) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 2 (2)
Chlamydial infection (Infections and infestations) | 12 (12) | 10 (10)
Urethritis chlamydial (Infections and infestations) | 6 (6) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 16 (19) | 2 (2)
Headache (Nervous system disorders) | 10 (10) | 8 (8)
Fatigue (General disorders) | 8 (9) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (8) | 0 (0)
Vision blurred (Eye disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT04010539/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT04010539/SAP_001.pdf